CLINICAL TRIAL: NCT01746121
Title: Clinical and Molecular Study of Amelogenesis Imperfecta
Brief Title: Amelogenesis Imperfecta
Status: Terminated | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4266
Record Dates: First submitted 2012-10-22; First posted 2012-12-10 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2013-02

CONDITIONS: Amelogenesis Imperfecta
MeSH Terms: conditions — Amelogenesis Imperfecta | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Amelogenesis Imperfecta: Salivary and blood sampling, as part of routine care. Collection of exfoliated teeth
  Interventions: Genetic: Salivary and blood sampling, as part of routine care. Collection of exfoliated teeth.
- healthy family members: Salivary and blood sampling, as part of routine care. Collection of exfoliated teeth
  Interventions: Genetic: Salivary and blood sampling, as part of routine care. Collection of exfoliated teeth.

INTERVENTIONS:
Genetic: Salivary and blood sampling, as part of routine care. Collection of exfoliated teeth.

SUMMARY:
Amelogenesis Imperfecta (AI) are a heterogeneous group of rare genetic diseases transmitted according to various mode of inheritance (X-linked, autosomal dominant, autosomal recessive) affecting the formation/mineralization of tooth enamel. These diseases exist in isolation with clinical manifestations limited to the oral cavity or may be associated to other symptoms in syndromes. Many different genes (AMELX, ENAM, ENAMELYSIN or MMP20, KLK4, DLX3, FAM83H, FAM20A WDR72…) coding for enamel matrix proteins, enamel matrix degrading proteins, proteins involved in hydroxyapatite formation and growth and mineralization processes have been discovered responsible for the clinical phenotypes (hypoplastic, hypomineralized, hypomature) encountered in AI.

Genes involved in enamel formation but not yet identified in association with any form of AI include: AMELY, AMELOBLASTIN, TUFTELIN, AMELOTIN, A Pin protein, ODAM (Odontogenic ameloblast associated).

In this research protocol the investigators explore the phenotype including the enamel ultrastructure and the genotype of a cohort of patients presenting AI.

ELIGIBILITY:
Inclusion criteria:

* Patient presenting with AI
* New patient or patient already known in the center
* Child (in his primary dentition) or adult
* Man or woman
* Having signed a consent form or accepted to participate to the study
* Patient affiliated to social security
* Validation of the inclusion by the principal investigator looking at the patient file

Exclusion criteria:

* Patient with acquired enamel defects
* Patient whose clinical diagnostic is not possible
* Patient whose clinical file does not contain teeth photos
* Patient who has not signed a consent form and accepted to participate to the study
* Patient who is not affiliated to social security.
* Non validation of the inclusion by the principal investigator looking at the patient file

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The recruitment of patients comes from several sources. A first cohort of 40 families is already followed by the reference center of Strasbourg. The reference center for rare diseases dental manifestations of Strasbourg recruiting patients at regional, interregional, national and international scale.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Natural history of Amelogenesis Imperfecta | at day of enrollment
  Familial, medical, dental history

SECONDARY OUTCOMES:
Phenotype of Amelogenesis Imperfecta | at day of enrollment
  Clinical and radiographic examination Type of enamel defects Associated dental or craniofacial anomalies

OTHER OUTCOMES:
Genetic Bases of Amelogenesis Imperfecta | within 3 years after enrollment
  Genetic analysis
Ultrastructure of teeth hard tissues | within 3 years after enrollment
  Ultrastructure analysis of teeth hard tissues

CONTACTS AND LOCATIONS:
Overall Officials: Bloch-Zupan Agnes, DChD, PhD, HDR, PU-PH, Principal Investigator — University Hospital of Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace, France

REFERENCES:
- [Derived] Bloch-Zupan A, Rey T, Jimenez-Armijo A, Kawczynski M, Kharouf N; O-Rare consortium; Dure-Molla M, Noirrit E, Hernandez M, Joseph-Beaudin C, Lopez S, Tardieu C, Thivichon-Prince B; ERN Cranio Consortium; Dostalova T, Macek M Jr; International Consortium; Alloussi ME, Qebibo L, Morkmued S, Pungchanchaikul P, Orellana BU, Maniere MC, Gerard B, Bugueno IM, Laugel-Haushalter V. Amelogenesis imperfecta: Next-generation sequencing sheds light on Witkop's classification. Front Physiol. 2023 May 9;14:1130175. doi: 10.3389/fphys.2023.1130175. eCollection 2023. PMID 37228816
- [Derived] Prasad MK, Geoffroy V, Vicaire S, Jost B, Dumas M, Le Gras S, Switala M, Gasse B, Laugel-Haushalter V, Paschaki M, Leheup B, Droz D, Dalstein A, Loing A, Grollemund B, Muller-Bolla M, Lopez-Cazaux S, Minoux M, Jung S, Obry F, Vogt V, Davideau JL, Davit-Beal T, Kaiser AS, Moog U, Richard B, Morrier JJ, Duprez JP, Odent S, Bailleul-Forestier I, Rousset MM, Merametdijan L, Toutain A, Joseph C, Giuliano F, Dahlet JC, Courval A, El Alloussi M, Laouina S, Soskin S, Guffon N, Dieux A, Doray B, Feierabend S, Ginglinger E, Fournier B, de la Dure Molla M, Alembik Y, Tardieu C, Clauss F, Berdal A, Stoetzel C, Maniere MC, Dollfus H, Bloch-Zupan A. A targeted next-generation sequencing assay for the molecular diagnosis of genetic disorders with orodental involvement. J Med Genet. 2016 Feb;53(2):98-110. doi: 10.1136/jmedgenet-2015-103302. Epub 2015 Oct 26. PMID 26502894